CLINICAL TRIAL: NCT05072652
Title: Short-term Immobilization and Rehabilitation of the Lower Limb: Changes in Strength, Size, and Neuromuscular Function
Brief Title: Short Term Immobilization of the Lower Limb
Acronym: STILL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Matt Stock, Associate Professor of Physical Therapy, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00003289
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Weakness, Muscle; Muscle Weakness; Muscle Loss; Muscle Atrophy; Injury, Knee
Keywords: immobilization; muscle atrophy; muscle strength; action observation; mental imagery; neuromuscular electrical stimulation; rehabilitation
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy; Knee Injuries

STUDY DESIGN:
Intervention Model Description: Repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immobilization (Experimental): Participants in the immobilization groups will undergo one week of unilateral knee joint immobilization of the left leg.
  Interventions: Other: Neuromuscular Electrical Stimulation; Other: Action Observation + Mental Imagery
- Control (No Intervention): The control group will not undergo any intervention.

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation — Participants in this group will perform twice daily neuromuscular electrical stimulation training sessions of the quadriceps muscles (specifically, the vastus lateralis and rectus femoris) or the immobilized left leg.
  Arms: Immobilization
Other: Action Observation + Mental Imagery — Participants in this group will perform daily action observation + mental imagery training via video and audio recordings.
  Arms: Immobilization

SUMMARY:
The purpose of this study is to determine the effects of one week of knee-joint immobilization on muscle size, strength, neuromuscular function, and brain function. In addition, the effects of two different interventions (i.e., neuromuscular electrical stimulation and action observation/mental imagery) throughout immobilization will be determined. Following the immobilization period, participants that have lost strength will be rehabilitated with twice weekly resistance training sessions, and sex-based differences in rehabilitation timelines will be examined.

DETAILED DESCRIPTION:
This study will utilize a repeated measures design in healthy adults aged 18-40 years. After a thorough familiarization visit, muscular size, strength, neuromuscular responses, and corticospinal excitability/inhibition will be measured before (PRE) and after (POST) one week of unilateral knee joint immobilization of the left leg. Four groups will be examined: 1) immobilization only, 2) immobilization + daily neuromuscular electrical stimulation, 3) immobilization + daily action observation/mental imagery training, 4) a control group. Throughout the immobilization period, participants will be in a leg brace locked at 90 degrees knee flexion. They will perform daily range of motion exercises and wear a compression sock at all times to mitigate the risk of blood clots. Following completion of the immobilization period, participants that have lost strength will complete a supervised rehabilitation program of twice weekly lower body resistance training sessions until they have returned to baseline levels of strength. Group assignment will be randomized and blocked on sex to ensure an equal number of participants within each group consisting of a relatively equal number of males and females.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between the ages of 18-40 years
* Body mass index >20 kg/m2 or < 35 kg/m2

Exclusion Criteria:

* Body mass index <20 kg/m2 or > 35 c
* Experience of major joint pain/discomfort of the upper or lower limbs, back, or neck within the previous six months.
* History of major musculoskeletal injury or surgery
* Neuromuscular disease (e.g., Parkinson's, MS, ALS)
* Metabolic disease (e.g., diabetes, thyroid disorder, metabolic syndrome)
* Personal or family history of blood clots
* Trouble using or controlling one's muscles
* History of cancer
* History of stroke
* History of heart attack
* History of arthritis
* Use of an assistive walking device or mobility aids within the past six months
* Use of anabolic steroids within the past six months
* History of convulsions, seizures, or syncope
* History of concussion as diagnosed by a physician
* Certain medications (e.g., muscle relaxants, benzodiazepines)
* Very thick hair or certain hairstyles that would impede the TMS coil from making direct contact with the scalp
* Allergy to rubbing alcohol
* Lack of transportation to and from the laboratory
* Implant of any kind
* Pregnancy
* Allergy to silver
* Diagnosis of any psychiatric condition

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants enrolled in this study must self identify with their biological sex at birth
Enrollment: 50 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Muscular strength | 15 minutes
  Changes in muscular strength will be measured via maximal voluntary contraction torque
Muscular size | 10 minutes
  Changes in muscular size will be measured via ultrasonography of the quadriceps
Corticospinal responses | 30 minutes
  Corticospinal responses will be measured with transcranial magnetic stimulation targeting the lower limbs
Motor unit behavior | 10 minutes
  Motor unit recruitment threshold and firing rate will be measured with surface electromyography signals detected from the quadriceps
Voluntary activation | 15 minutes
  Voluntary activation will be measured using the interpolated twitch technique
Rate of recovery | 1.5 hours per session
  The time taken to recover strength lost will be measured via number of resistance training sessions needed after immobilization

SECONDARY OUTCOMES:
Compliance | one week
  Compliance will be measured via the use of accelerometers around both ankles. Compliance will be calculated as the number of participants that following the crutch/brace protocol as described.
Physical activity (Step count) | one week
  Physical activity will be assessed via step counts and compared to changes in primary outcome measures via accelerometers around both ankles

CONTACTS AND LOCATIONS:
Overall Officials: Matt S Stock, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared by the PI upon reasonable request. Personal identifiable information will not be shared; however, physiological data and outcome measures may be shared if requested.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available upon reasonable request after the time of study completion and manuscript publication
Access Criteria: To access IPD, please contact the study PI.

REFERENCES:
- [Derived] Harmon KK, Girts RM, Rodriguez G, Beausejour JP, Pagan JI, Carr JC, Garcia J, Roberts MD, Hahs-Vaughn DL, Stout JR, Fukuda DH, Stock MS. Combined action observation and mental imagery versus neuromuscular electrical stimulation as novel therapeutics during short-term knee immobilization. Exp Physiol. 2024 Jul;109(7):1145-1162. doi: 10.1113/EP091827. Epub 2024 Apr 30. PMID 38687158
- See also: Related Info — https://healthprofessions.ucf.edu/research/studies/